CLINICAL TRIAL: NCT07338565
Title: Magnesium Status in Patients With Gastrointestinal Disease
Brief Title: Magnesium in Gastrointestinal Disease
Acronym: MAGIC
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Steno Diabetes Center Aarhus, Denmark (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-41-25
Record Dates: First submitted 2025-11-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Colitis Ulcerosa; Colitis Ulcerative; Crohns Disease; Morbus Crohn; Ileostomy - Stoma; Ileostoma; Ileostomies; Bile Acid Diarrhea; Bile Acid Malabsorption; Magnesium Deficiency; Magnesium Level; Magnesium
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Magnesium Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMC), buffy coat, red blood cells, muscle tissue, and intestinal mucosal biopsies (optional) will be retained for analysis of magnesium and related biomarkers. Although not intended for genetic testing, these samples contain genomic DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with an gastorintestinal disease or conditions: Patients with inflammatory bowel disease, ileostomy or bile acid diarrhoea
- Healthy individuals (control group): Healthy individuals (control group)

SUMMARY:
Individuals with gastrointestinal diseases - such as Crohn's disease, ulcerative colitis, ileostomy, or bile acid diarrhoea - are at increased risk of magnesium deficiency. Magnesium is a vital mineral that supports many essential functions in the body, including muscle contraction, nerve signalling, heart rhythm, and bone health. Deficiency may contribute to fatigue, muscle cramps, abnormal heart rhythms, and reduce the quality of life.

The purpose of this study is to investigate the prevalence of magnesium deficiency in individuals with these conditions and to identify the most accurate and practical methods for assessing magnesium status in clinical care.

Although plasma magnesium is commonly used in routine blood tests, it represents only about 1% of the body's total magnesium and may not reflect true magnesium levels within cells or tissues. Hence, this study compares several different ways of measuring magnesium, including:

* Plasma magnesium
* Magnesium levels in red and white blood cells (PBMC, RBC, and buffy coat)
* Magnesium levels in muscle tissue (via biopsy)
* A magnesium retention test, based on how much magnesium is excreted after an infusion

The study includes four groups:

1. Patients with inflammatory bowel disease.
2. Patients with an ileostomy.
3. Patients with bile acid diarrhoea.
4. Healthy individuals (control group).

All participants will provide blood and urine samples, and some may undergo optional biopsies of muscle or intestinal tissue. Participants will also complete questionnaires and undergo tests of muscle strength and body composition.

The findings are expected to enhance the understanding and detection of magnesium deficiency in patients with gastrointestinal diseases and to aid in the development of more effective tools for identifying and treating this common yet often overlooked condition.

DETAILED DESCRIPTION:
This cross-sectional study aims to improve the assessment of magnesium status in patients with chronic intestinal diseases. The study will evaluate and compare a range of biochemical and functional markers to determine which provide the most accurate, reliable, and clinically useful reflection of whole-body magnesium status. The long-term goal is to support the development of a more sensitive screening strategy for magnesium deficiency in clinical practice, especially for populations at increased risk due to gastrointestinal losses or malabsorption.

Magnesium deficiency is often underdiagnosed due to the limitations of standard plasma magnesium measurement. Although total body magnesium is primarily stored in bone and soft tissue, the current standard diagnostic method (plasma magnesium) reflects only a small fraction of total magnesium (<1%) and does not correlate well with intracellular magnesium content. As a result, many cases of subclinical or functional magnesium deficiency go undetected, particularly in populations with chronic gastrointestinal conditions that alter absorption and excretion.

Study Design and Rationale:

The study will consist of four visits and include two groups:

1. Patients with gastrointestinal disease or conditions, divided into three subgroups: those with inflammatory bowel disease (IBD; Crohn's disease or ulcerative colitis), those with an ileostomy or patients with bile acid diarrhoea.
2. Healthy controls without known gastrointestinal disease.

The three patient subgroups are selected based on known risk factors for magnesium depletion: chronic diarrhoea, intestinal resection, and malabsorption. The healthy control group serves as a reference population.

All participants will undergo a standardised clinical examination and biological sampling protocol, including:

* Blood sampling for plasma magnesium, ionised magnesium, and intracellular magnesium (PBMC, RBC, and buffy coat)
* 24-hour urine collection for magnesium excretion
* An intravenous magnesium loading test (retention test)
* Muscle biopsy for quantification of total magnesium concentration in skeletal muscle
* Faecal sample for analysis of gut microbiome composition
* Assessment of muscle function (handgrip strength test and sit-to-stand test)
* Body composition measurement (bioimpedance analysis)
* Patient reporting outcomes covering fatigue, gastrointestinal symptoms, mental well-being, and quality of life
* Food frequency questionnaire assessing dietary magnesium intake

A subset of participants undergoing clinically indicated endoscopic procedures will have intestinal biopsies (duodenal or colonic mucosa) collected for exploratory analyses of tissue magnesium concentration and expression of magnesium transporters, including TRPM6, TRPM7, CNNM4, and SLC41A1.

Analytical Methods:

Magnesium concentrations will be measured using inductively coupled plasma mass spectrometry (ICP-MS), which allows for highly sensitive and specific quantification of total magnesium content in various biological matrices. Plasma and urine samples will be analysed for total magnesium and ionised magnesium, where applicable.

Intracellular magnesium in peripheral blood mononuclear cells (PBMCs), red blood cells (RBCs), and buffy coat will be analysed following standardised separation protocols. Special precautions are taken during sample handling and storage to avoid trace metal contamination, including the use of trace metal-free collection tubes, ultrapure reagents, and certified laboratory plastics.

Muscle tissue samples will be cryopreserved and analysed in collaboration with a reference laboratory with expertise in trace metal tissue analysis. Before digestion and ICP-MS quantification, tissue samples may undergo lyophilisation and homogenization under clean-room conditions.

For participants completing the magnesium retention test, baseline urinary magnesium excretion will be compared to excretion after a standardised intravenous magnesium sulfate load. Magnesium retention will be calculated as the difference between the infused magnesium dose and the amount excreted in urine during 24 hours. This method is regarded as the reference standard for assessing total body magnesium stores, but is rarely used in clinical practice due to its complexity.

Data Handling and Statistical Analysis:

Data will be collected using REDCap and stored on secure institutional servers with access restricted to study personnel. All participants will be assigned a unique study ID to ensure confidentiality. Descriptive statistics will be used to summarise demographic and clinical characteristics. Differences between groups will be analysed using appropriate statistical tests (e.g., ANOVA, Kruskal-Wallis, chi-square) depending on data distribution.

Correlation analyses will be performed to compare plasma magnesium with intracellular and tissue magnesium levels. Receiver Operating Characteristic (ROC) curves may be generated to evaluate the sensitivity and specificity of various biomarkers against the magnesium retention test and/or muscle magnesium content as reference standards.

Subgroup analyses may explore differences based on disease type, presence of resection, disease activity, medication use (e.g., proton pump inhibitors, diuretics), and nutritional intake.

Ethical Considerations:

The study has been reviewed and accepted by the relevant Research Ethics Committee and complies with the Declaration of Helsinki and national legislation on research ethics. Written informed consent will be obtained from all participants before any study procedures. Muscle biopsy and intestinal biopsy are optional and only performed in participants who consent to these procedures.

Participants are informed of potential risks related to muscle biopsy (e.g., bruising, soreness, rare risk of infection) and intravenous magnesium infusion (e.g., transient warmth, flushing, hypotension). All biological samples will be stored and handled under current regulations for biobank material and may be used for future research within the same scope if participants provide consent.

Expected Impact:

This study is expected to provide new insights into the clinical evaluation of magnesium status in patients with gastrointestinal diseases. By comparing traditional and alternative markers of magnesium status with reference measures such as muscle magnesium and magnesium retention, the study will help identify more accurate, practical, and scalable methods for detecting deficiency in at-risk populations.

The findings may inform future guidelines on nutritional screening, support earlier diagnosis of magnesium deficiency, and contribute to improved management of symptoms and comorbidities related to chronic magnesium depletion.

ELIGIBILITY:
Inclusion Criteria:

- Age 18 or older, mentally competent, and able to understand Danish.

Group 1:

- Diagnosed with IBD (DK50X, Crohn's disease, or DK51X, ulcerative colitis), ileostomy (DZ932) or bile acid diarrhoea (DSK908B) (Se-HCAT scintigraphy showing residual activity <10%).

Group 2:

- Healthy individuals.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Use of oral magnesium supplements for more than 2 weeks before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will primarily be recruited from both inpatient and outpatient clinics from the Department of Hepatology and Gastroenterology at Aarhus University Hospital, as well as through patient associations (Colitis-Crohn Association and the Danish Stoma Association). Healthy individuals will be recruited through online platforms/social media and local hospital networks.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with magnesium deficiency (magnesium retention >20%) | Immediately after completion of the magnesium infusion (Visit 3; urine collection completed within ~24 hours post-infusion).
  Proportion of participants whose magnesium retention rate exceeds 20%, where retention (%) = (infused magnesium - urinary magnesium excretion) / infused magnesium × 100.
  Unit: percent (%). Threshold for deficiency: retention >20%.

SECONDARY OUTCOMES:
PBMC magnesium concentration | Through study completion, an average of 5 weeks.
  Total magnesium concentration in peripheral blood mononuclear cells (PBMC). Units: nmol/10⁶ cells.
RBC magnesium concentration | Through study completion, an average of 5 weeks.
  Magnesium concentration in red blood cells (RBC). Units: nmol/10⁶ cells.
Buffy coat magnesium concentration | Through study completion, an average of 5 weeks.
  Total magnesium concentration in the buffy coat fraction. Units: nmol/10⁶ cells.
Intraindividual variability of PBMC magnesium (coefficient of variation) | Through study completion, an average of 5 weeks.
  Within-subject coefficient of variation (CV%) for PBMC magnesium
Intraindividual variability of RBC magnesium (coefficient of variation) | Through study completion, an average of 5 weeks.
  Within-subject coefficient of variation (CV%) for RBC magnesium
Intraindividual variability of buffy coat magnesium (coefficient of variation) | Through study completion, an average of 5 weeks.
  Within-subject coefficient of variation (CV%) for buffy coat magnesium.
24-hour urinary magnesium excretion (mmol/day) | Through study completion, an average of 5 weeks.
  Total magnesium excreted in 24-hour urine collection, expressed in millimoles per 24 hours (mmol/24 h).
Skeletal muscle magnesium concentration | Visit 1 (Baseline).
  Intracellular magnesium concentration measured in skeletal muscle biopsy tissue, expressed as mmol per kg.
Gut microbiota composition (relative abundance) | Visit 1 (Baseline)
  Taxonomic composition and diversity metrics (alpha and beta diversity) from 16S/shotgun sequencing; reported as relative abundance (%) and diversity indices (unitless).
Bone mineral density (BMD) by DEXA (g/cm²) | Visit 1 (Baseline).
  Units = grams per square centimetre (g/cm²).
Plasma metabolic markers | Visit 1 (Baseline), Visit 2 (Day 2), Visit 3 (Day 3), and Visit 4 (end of study; 4 weeks after Visit 3).
  Mean plasma glucose (HbA1c, mmol/mol)
Maximum handgrip strength (kg) | Visit 1 (Baseline).
  Maximal isometric grip strength is measured by a calibrated dynamometer in kilograms (kg). If multiple attempts, report the best of three. Higher = greater strength.
SIBDQ score - Short Inflammatory Bowel Disease Questionnaire (10-70) | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  Total SIBDQ score from 10 (worst) to 70 (best); higher values indicate better quality of life.
Estimated daily magnesium intake (MgFFQ) (mg/day) | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  Estimated magnesium intake derived from the Magnesium Food Frequency Questionnaire (MgFFQ), reported in mg/day.
Magnesium concentration in intestinal tissue | Visit 1 (Baseline).
  Unit: mmol/kg.
Plasma hormonal markers | Visit 1 (Baseline), Visit 2 (Day 2), Visit 3 (Day 3) and Visit 4 (end of study; 4 weeks after Visit 3)
  Fasting plasma insulin, plasma parathyroid hormone (PTH). Unit: pmol/L
Plasma creatinine | Visit 1 (Baseline), Visit 2 (Day 2), Visit 3 (Day 3) and Visit 4 (end of study; 4 weeks after Visit 3)
  Plasma creatinine (µmol/L)
Plasma inflammatory marker | Visit 1 (Baseline), Visit 2 (Day 2), Visit 3 (Day 3) and Visit 4 (end of study; 4 weeks after Visit 3)
  Plasma C-reactive protein (CRP, mg/L)
Plasma Renin | Visit 1 (Baseline), Visit 2 (Day 2), Visit 3 (Day 3) and Visit 4 (end of study; 4 weeks after Visit 3)
  Unit: × 10-³ IU/L
Plasma Aldosterone | Visit 1 (Baseline), Visit 2 (Day 2), Visit 3 (Day 3) and Visit 4 (end of study; 4 weeks after Visit 3)
  Unit: pmol/l
Leukocyte differential count | Visit 1 (Baseline), Visit 2 (Day 2), Visit 3 (Day 3) and Visit 4 (end of study; 4 weeks after Visit 3)
  Unit: 10⁹/L
Urinary creatinine | Visit 2 (Day 2) and Visit 3 (Day 3)
  24-hour urinary creatinine (mmol/day)
Urine volume | Visit 2 (Day 2) and Visit 3 (Day 3)
  24-hour urine volume (mL/day)
24-hour urinary acid-base excretion (mmol/day) | Visit 2 (Day 2)
  Net acid excretion and components (ammonium, titratable acids) from 24-hour urine, reported in mmol/day.
Creatinine clearance | Visit 2 (Day 2) and Visit 3 (Day 3)
  Unit = mL/min)
Faecal bicarbonate concentration | Visit 1 (Baseline).
  Unit = mmol/L
Bone mineral content (BMC) by DEXA (g) | Visit 1 (Baseline).
  BMC in grams measured by DEXA.
Appendicular lean mass (ALM) (kg) | Visit 1 (Baseline).
  Sum of lean mass of arms and legs measured by DEXA, reported in kilograms (kg).
Total lean mass by DEXA (kg) | Visit 1 (Baseline).
  Whole-body lean mass in kg.
Total fat mass by DEXA (kg) | Visit 1 (Baseline).
  Whole-body fat mass in kg.
BIS Resistance (R, Ω) | Visit 1 (Baseline).
  Bioimpedance spectroscopy resistance measured at specified frequencies, reported in ohms (Ω).
30-second Sit-to-Stand test (repetitions) | Visit 1 (Baseline).
  Number of full stands completed in 30 seconds. Higher = better lower-body function.
BIS Reactance (Xc, Ω) | Visit 1 (Baseline).
  Bioimpedance reactance in ohms (Ω).
Phase angle (degrees) by BIS (°) | Visit 1 (Baseline).
  Phase angle derived from BIS, in degrees. Higher values generally indicate better cell integrity.
Total Body Water (TBW), Intracellular Water (ICW) and Extracellular Water (ECW) (liters) | Visit 1 (Baseline).
  Body water compartments measured by BIS or D₂O, reported in litres (L). ECW/ICW ratio also to be reported (unitless).
SBS-QoL score - Short Bowel Syndrome Quality of Life (0-100) | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  Total score from 0 to 100; higher indicates better quality of life. State whether raw or normalized score used.
EQ-5D-5L index value. | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  EQ-5D-5L index score (range typically from <0 to 1); higher indicates better health.
IBD-Fatigue Scale total score (specify range used) | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  IBD-Fatigue Scale total score (specify instrument range, e.g., 0-100); higher = greater fatigue.
Harvey-Bradshaw Index (HBI) total score (Crohn's disease activity) | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  HBI total score (range 0->16); higher = more severe disease activity.
Simple Clinical Colitis Activity Index (SCCAI) total score | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  SCCAI total score (range 0-19); higher = worse ulcerative colitis activity.
Visual analogue scale (VAS) for magnesium-deficiency symptoms (0-100 mm) | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  Participant-reported symptom severity on 100-mm VAS; 0 = no symptom, 100 = worst possible symptom. Higher = worse.
KRAM questionnaire composite scores (diet, smoking, alcohol, physical activity) | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  KRAM domains scored per instrument instructions; report component scores (units as instrument defines).
Intestinal tissue magnesium concentration | Visit 1 (Baseline).
  Magnesium content measured in intestinal mucosal biopsy tissue expressed as mmol per kg.
Plasma electrolytes (mmol/L) | Through study completion, an average of 5 weeks.
  Plasma concentrations of magnesium, calcium, sodium and potassium, each expressed in millimoles per litre (mmol/L).
  Individual analytes are reported separately under this grouped title.
Fasting plasma glucose (mmol/L) | Visit 1 (Baseline) and Visit 4 (end of study; 4 weeks after Visit 3).
  Fasting plasma glucose measured in mmol/L.
Plasma albumin (g/L) | Through study completion, an average of 5 weeks.
  Plasma albumin concentration in grams per liter (g/L).
Spot urine magnesium concentration (mmol/L) | Visit 2 (Day 2) and Visit 3 (Day 3)
  Magnesium concentration in a single spot urine sample, expressed as millimoles per litre (mmol/L).
24-hour urinary creatinine | Visit 2 (Day 2) and Visit 3 (Day 3)
  Creatinine excretion measured in 24-hour urine (mmol/day). Used to verify completeness of the collection.
Spot urine acid-base parameters | Visit 2 (Day 2) and Visit 3 (Day 3)
  Acid-base markers in spot urine (e.g., NH₄⁺, titratable acids) expressed in mmol/L.
Serum acid-base status: bicarbonate, base excess, total CO₂ | Visit 1 (Baseline).
  Arterial/venous serum pH, bicarbonate (mmol/L), base excess (mmol/L) and total CO₂.
  Unit: mmol/L.
Estimated glomerular filtration rate (eGFR, mL/min/1.73 m²) | Visit 1 (Baseline).
  eGFR calculated using CKD-EPI formula (or local lab algorithm), reported in mL/min/1.73 m².

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus N, Denmark